CLINICAL TRIAL: NCT05923151
Title: Techniques and Advantages of the Cranial-caudal Mixed Medial Approach for Laparoscopic Right Hemicolectomy With Complete Mesocolic Excision
Brief Title: The Cranial-caudal Mixed Medial Approach for Laparoscopic Right Hemicolectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jie Wang (Other)
Collaborators: Yangzhou University (Other)
Responsible Party: Sponsor-Investigator, Jie Wang, Principal Investigator, Subei People's Hospital of Jiangsu Province
Organization: Subei People's Hospital of Jiangsu Province (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SubeiH
Record Dates: First submitted 2023-06-09; First posted 2023-06-28 (Actual); Last update posted 2023-06-28 (Actual); Status verified 2023-06

CONDITIONS: Intraoperative Blood Loss; Postoperative Complications; Pathology
MeSH Terms: conditions — Postoperative Complications

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The cranial-caudal mixed medial approach group (Experimental): 75 patients were diagnosed with right colon cancer and underwent the cranial-caudal mixed medial approach for laparoscopic right hemicolectomy with complete mesocolic excision.
  Interventions: Procedure: The cranial-caudal mixed medial approach
- the medial approach group (Other): 73 patients were diagnosed with right colon cancer and underwent the medial approach for laparoscopic right hemicolectomy with complete mesocolic excision.
  Interventions: Procedure: The cranial-caudal mixed medial approach

INTERVENTIONS:
Procedure: The cranial-caudal mixed medial approach — Expose the fusion fascia of Transverse colon mesocolon and stomach, and cut the gastrocolic ligament. The mesentery of Transverse colon was dissociated from the medial side to the lateral side along the gastroepiploic vessels to expose the branches of Henle's trunk and the right colon vessels. The dorsal mesentery of the small intestine is cut along the "yellow white line", and free cephalically along the Toldt space to separate the posterior space of the Ascending colon and the anterior space of the pancreas and duodenum behind the Transverse colon. The right colon blood vessels were dissected along SMV from the projection of ileocolic blood vessels, and the blood vessels were cut off by high ligation, and the lymph nodes at the root of Mesentery were cleared. Through a small incision in the middle of the abdomen, the right colon and mesentery were completely removed to complete digestive tract reconstruction.

SUMMARY:
To explore the feasibility and effectiveness of the cranial-caudal mixed medial approach in laparoscopic right hemicolectomy with complete mesocolic excision. Laparoscopic right hemicolectomy using the cranial-caudal mixed medial approach is safe and feasible, can shorten the operation time, reduce the risk of intraoperative bleeding, and has good clinical results.

DETAILED DESCRIPTION:
The data of patients undergoing laparoscopic right hemicolectomy performed in the same surgical group of gastrointestinal surgery at Northern Jiangsu People's Hospital from February 2017 to June 2022 were retrospectively analyzed. According to different surgical approaches, patients were divided into the cranial-caudal mixed medial approach group and the medial approach group.

Intraoperative and postoperative data were collected. Intraoperative data is obtained through surgical records and pathological reports, including total operation time, Laparoscopic procedure time, Intraoperative blood loss, sample length, number of lymph nodes collected, and number of positive lymph nodes. Postoperative data includes exhaust time, liquid intake time, postoperative hospitalization and complications. Among them, complications are short-term postoperative complications (surgical related complications, non-surgical related complications) within the first 30 days after surgery (or throughout the hospitalization period, if more than 30 days, and are classified according to the Clavien-Dindo classification method.

To explore the feasibility and effectiveness of the cranial-caudal mixed medial approach in laparoscopic right hemicolectomy with complete mesocolic excision.

ELIGIBILITY:
Inclusion Criteria:

* Age range: 18-70 years old
* Right colon cancer confirmed by colonoscopy and pathological diagnosis
* Single primary tumor without distal metastasis
* Laparoscopic operation

Exclusion Criteria:

* Age below 18 and above 70 years old
* Patients who need urgent surgery
* Persons with a history of malignant tumors
* Multiple primary tumors or distant metastases

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 148 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2023-02-01 (Actual)

PRIMARY OUTCOMES:
The operative time | Surgery start (skin incision time) - Surgery end (suture incision end time)
  The length of operative time

SECONDARY OUTCOMES:
Intraoperative blood loss | Surgery start (skin incision time) - Surgery end (suture incision end time)
  Measurement by gauze transfusion weighing method: soaked 32cm × A 20cm sized gauze loses approximately 30ml of blood; Soak 36cm × A 36cm sized gauze loses approximately 50ml of blood.

OTHER OUTCOMES:
Number of lymph nodes cleaned | 3-5 days after surgery
  Number of lymph node dissection
Anastomotic leakage | Within 30 days after surgery
  Positive bacterial culture in peritoneal drainage fluid
Liver failure | Within 30 days after surgery
  ASL and ALT indicators in liver function examination
Renal failure | Within 30 days after surgery
  BUN and Cr indicators in renal function examination

CONTACTS AND LOCATIONS:
Locations (1):
- Subei People's Hospital, Yangzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No